CLINICAL TRIAL: NCT05494242
Title: Single Superior Internal Limiting Membrane/Epiretinal Membrane Flap for the Full Thickness Macular Hole
Brief Title: Single Superior ILM/ERM Flap for the FTMH.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omer Othman Abdullah (Other)
Collaborators: Ibinsina Modern Eye and Retina Center (Other)
Responsible Party: Sponsor-Investigator, Omer Othman Abdullah, Associate consultant ophthalmologist, Ibinsina Modern Eye and Retina Center
Organization: Ibinsina Modern Eye and Retina Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IMER 99
Record Dates: First submitted 2022-08-06; First posted 2022-08-09 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Ophthalmopathy
Keywords: Full thickness macular hole; Epiretinal membrane; Internal limiting membrane; Flap
MeSH Terms: conditions — Eye Diseases; Epiretinal Membrane | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- single superior flap technique to secure macular hole closure. (Experimental): The patients are divided into two groups:
  For the first group, the flap will be carried out under the effect of perfluorocarbon.
  For the second group, the flap stabilized with methylcellulose.
  Interventions: Other: Surgical intervention
- Double flap technique to secure macular hole closure. (Active Comparator): This arm is NCT05269563, we utilize the results as a comparator to the superior single flap technique.
  Interventions: Other: Surgical intervention

INTERVENTIONS:
Other: Surgical intervention — Pars-plana vitrectomy.

SUMMARY:
In this study, the investigators will make the only upper flap either from the internal limiting membrane or from the epiretinal membrane to cover the full thickness macular hole.

DETAILED DESCRIPTION:
After the investigators completed the clinical trial NCT05269563, which was a double flap technique; that consists of two flaps from the internal limiting membrane and the epiretinal membrane. The inferior flap was implanted inside the hole, but the upper flap was utilized to cover the hole. The results were encouraging. Therefore, in this study, the investigators will make the only upper flap to cover the full thickness macular hole, to compare both visual and anatomical outcomes with the double flapped technique (NCT05269563) results. Therefore the double flap will be our control.

ELIGIBILITY:
Inclusion Criteria:

* Full thickness macular hole

Exclusion Criteria:

* Lamellar and pseudo holes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-03-21 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Anatomical outcome | The fourth weeks post-operatively
  OCT

SECONDARY OUTCOMES:
Functional outcome | The fourth week post-operatively.
  Best corrected visual acuity

CONTACTS AND LOCATIONS:
Locations (1):
- Omer Othman Abdullah, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: Yes
Both the best corrected visual acuity and the OCT.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Expected to be available around the end of November 2022
Access Criteria: via your permisson